CLINICAL TRIAL: NCT06433167
Title: Investigation of Gait Pattern in Idiopathic Scoliosis
Status: Not yet recruiting | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, İnci Hazal Ayas, Research asistant, Gazi University
Other Study IDs: Iayas9
Record Dates: First submitted 2024-05-18; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Idiopathic Scoliosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Idiopathic Scoliosis: The patient group for this research comprises patients diagnosed with idiopathic scoliosis, a condition characterized by abnormal lateral curvature of the spine of unknown cause.
  Interventions: Other: Pedobarographic analysis
- Healthy control: Healthy control group is healthy individuals without any diagnosed disease.
  Interventions: Other: Pedobarographic analysis

INTERVENTIONS:
Other: Pedobarographic analysis — During the pedobarographic analysis, the patient takes steps on the platform at a regular walking speed, with arms relaxed at the sides, following a natural gait. In static analysis, measurements are taken while the patient remains stationary on the platform with arms in a relaxed position beside the body. Five measurements are separately recorded for both feet during the phases of stepping, heel strike, and toe lift. These measurements capture the highest pressures on the back of the foot, the middle part of the foot, and the inner, middle, and lateral sides of the front of the foot, including the toes. The pressure, force, and pressure-time integral corresponding to each area are then used to determine how and for how long these areas are exposed to pressure.

SUMMARY:
Scoliosis is a condition characterized by an abnormal curvature of the spine, which can affect an individual's gait. Scoliosis can alter body balance and weight distribution. Pedobarographic analysis identifies imbalances and abnormal pressure points by measuring the distribution of pressure applied to the sole of the foot. This examination helps detect abnormalities in the gait mechanics of individuals with scoliosis. Gait analysis can identify long-term foot and leg problems caused by scoliosis at an early stage, allowing for early interventions to prevent more serious issues.

The aim of this study is to analyze gait in individuals with idiopathic scoliosis and compare it with that of healthy individuals. The study will include 30 scoliosis patients who visited the Department of Orthopedics and Traumatology at Gazi University Hospital and were diagnosed with idiopathic scoliosis by a specialist physician. The gait patterns of the patients will be evaluated using pedobarography. Information about the type and degree of scoliosis will be obtained from hospital records. The results of this study may provide an objective and detailed evaluation of gait and pressure distribution disorders in individuals with scoliosis and may contribute to more effective treatment plans.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic scoliosis by an orthopedist
* The Cobb angle measured on the standard scoliosis radiograph should fall within the range of 10°-45°.

Exclusion Criteria:

* Presence of any orthopedic or neurological disease affecting trunk and extremity mobility, excluding scoliosis.
* History of previous spine or orthopedic surgery.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will include 30 scoliosis patients who visited the Department of Orthopedics and Traumatology at Gazi University Hospital and were diagnosed with idiopathic scoliosis by a specialist physician and 30 healty control without scoliosis.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Pedobarography | Day 1
  This assessment uses a specialized device called a pedobarograph, which consists of pressure sensors embedded in a platform. When a person stands or walks on the pedobarograph, the sensors record the pressure exerted by different parts of the foot. The resulting data is then used to create detailed pressure maps and graphs that highlight areas of high and low pressure.

CONTACTS AND LOCATIONS:
Overall Officials: İnci H Ayas, Msc, Study Director — Gazi University; Furkan Aral, MD, Study Chair — Gazi University; Burak Oklaz, MD, Study Chair — Gazi University; Ulunay Kanatlı, MD, Principal Investigator — Gazi University
Locations (1):
- Gazi University Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No